CLINICAL TRIAL: NCT00290056
Title: Effect of Supplemental Intake of Omega-3 Polyunsaturated Fatty Acids on the Rate and Complexity of Spontaneously Occurring Ventricular and Supraventricular Arrhythmias in Patients With Implantable Cardioverter Defibrillator (ICD) - A Randomized Clinical Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dalit Weisman, Sheba Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SHEBA-04-3494-DL-CTIL
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Last update posted 2009-11-04 (Estimated); Status verified 2009-11

CONDITIONS: Coronary Artery Disease; Arrhythmia
Keywords: CHD; Arrhythmia; ICD; Omega-3 PUFA; Nutrition
MeSH Terms: conditions — Coronary Artery Disease; Arrhythmias, Cardiac | interventions — Eicosapentaenoic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Eicosapentanoic acid (EPA) and Docosahexanoic acid (DHA). — 3.6 gram oral supplementation for 6 months.

SUMMARY:
We hypothesize that oral supplementation with omega-3 PUFA will decrease occurrence of arrhythmic events among post-MI, ICD recipients.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, crossover, double- blind interventional study. Patients will receive 3.6 g of EPA and DHA fish oil and placebo oil for 6 months, randomly, in a crossover design, with a four month washout period between treatments.

Randomization will be stratified by ejection fraction (≤ 35% or > 35%), and the type of the index arrhythmia (VT - spontaneous or inducible by electrophysiologic study (EPS), versus other - VF, SCD, Primary prevention - MADIT II).

Ischemia severity was chosen to be evaluated by Single Photon Emission Computed Tomography (SPECT) during stress (dipyridamol infusion).

Subcutaneous adipose-tissue biopsy, a biomarker considered the gold-standard for the objective assessment of long-term habitual dietary intake of fish and marine omega-3 PUFA (EPA and DHA) will be obtain.

Compliance will be monitored by counting returned capsules or bottles and by measuring the omega-3 PUFA composition in red blood cells (RBC).

Three different types of questionnaires will be used in this trial to obtain more information as to the additional potential benefit of omega-3 PUFA supplementation:

1. The newly Israeli Food Frequency Questionnaire (FFQ) will be used to examine dietary intake of other nutritional habits/patterns and its relationship to the study outcomes.
2. The Hebrew language SF-36 health survey will be used to examine general health status.
3. The Back questionnaires will be use to examine possible beneficial effects of fish oil supplementation on depressive symptomatology.

ELIGIBILITY:
Inclusion Criteria:

* post-MI patients.
* Both single and Dual chamber ICD recipient.
* implanted more than 3 months ago.
* Agree to give written informed consent.

Exclusion Criteria:

* Less than 18 years of age.
* ICD implantation as a 'bridge' to heart transplantation.
* Stable antiarrhythmic medication over the last month prior to enrollment.
* Patients taking class I antiarrhythmic medication.
* A projected lifespan less than one year.
* Participation in another trial (during or within 90 days before the study).
* Use of supplemental n-3 fatty acids during the last 3 months.
* Women who are pregnant and of childbearing potential who do not use adequate contraception.
* Patients known to have a history of recent drug or alcohol abuse. 10) History or current intestinal or hepatic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2005-11; Primary Completion 2009-11 (Actual); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
number of VT/VF episodes | continous

SECONDARY OUTCOMES:
All-cause mortality, cardiac mortality, recurrent and myocardial infarction. | continous
Atrial arrhythmia and non-sustained ventricular arrhythmia (non-sustained VT or ventricular premature complex (PVC)) as documented by ICD memory or 24 hour ECG (Holter) recording. | 24 hours
Whether omega-3 PUFA supplementation exerts different effects according to ischemia severity assessed by stress perfusion nuclear imaging. | time of the test

CONTACTS AND LOCATIONS:
Overall Officials: David Luria, MD, Principal Investigator — Sheba Medical Center
Locations (2):
- Israel (2):
  - The Tel Aviv Sourasky Medical Center, Tel Aviv
  - Sheba Medical Center, Heart Institute, Electrophysiology Unit, Tel Litwinsky